CLINICAL TRIAL: NCT04469998
Title: A Phase I/II, Randomized, Double-Masked, Vehicle-Controlled Study of the Safety, Tolerability, and Efficacy of AXR-270 Topical Eyelid Cream in Treating Posterior Blepharitis Associated With Meibomian Gland Dysfunction
Brief Title: Evaluation of AXR-270 for the Treatment of Posterior Blepharitis Associated With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AxeroVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXR201901
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Posterior Blepharitis; Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Posterior Blepharitis
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AXR-270 Low Dose (Experimental): AXR-270 Low Dose administered once daily
  Interventions: Drug: AXR-270 Low Dose
- AXR-270 High Dose (Experimental): AXR-270 High Dose administered once daily
  Interventions: Drug: AXR-270 High Dose
- AXR-270 Vehicle (Placebo Comparator): AXR-270 Vehicle administered once daily
  Interventions: Drug: AXR-270 Vehicle

INTERVENTIONS:
Drug: AXR-270 Low Dose — AXR-270 Topical Eyelid Cream
  Arms: AXR-270 Low Dose
Drug: AXR-270 High Dose — AXR-270 Topical Eyelid Cream
  Arms: AXR-270 High Dose
Drug: AXR-270 Vehicle — AXR-270 Topical Eyelid Cream Vehicle
  Arms: AXR-270 Vehicle

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of AXR-270 Cream in treating posterior blepharitis associated with Meibomian Gland Disease (MGD)

DETAILED DESCRIPTION:
AXR201901 is a multicenter, randomized, double-masked, vehicle-controlled study of AXR-270 cream and AXR-270 vehicle in subjects with signs and symptoms of posterior blepharitis associated with meibomian gland dysfunction

ELIGIBILITY:
Inclusion Criteria:

Male or female, 18 years or older

Have a clinical diagnosis of moderate to severe MGD (total MGD score between 5 and 14 on a scale with a range between 0 and 15; and clinical severity score of eyelid margin vascularity of at least 2 (moderate))

Have a score of ≥35 on Eye Discomfort using VAS

Have a tFCS score between 3 and 14 on the NEI scale

Have a Schirmer score of >7 mm

Have a OSDI score >30

If female, then subject should be non-pregnant and non-lactating

Exclusion Criteria:

Subjects with iritis, uveitis in either eye

Subjects with conjunctivitis, keratitis, severe anterior keratitis not related to MGD

Subjects with lid abnormalities

Subjects with ocular fungal, viral or bacterial infection

Subjects unable or unwilling to withhold the use of eyelid scrubs

Subjects with glaucoma and serious systemic disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Houman D Hemmati, MD, PhD, Study Director — AxeroVision, Inc.
Locations (1):
- AxeroVision, Inc., Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AXR-270 Low Dose: AXR-270 Low Dose administered once daily
  AXR-270 Low Dose: AXR-270 Topical Eyelid Cream 0.2%
- AXR-270 High Dose: AXR-270 High Dose administered once daily
  AXR-270 High Dose: AXR-270 Topical Eyelid Cream 2%
Period: Full Analysis Set (ITT Population)
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle
Started | 43 (One subject was randomized to AXR-270 Low Dose but received Vehicle instead) | 44 | 42 (One subject was randomized to AXR-270 Low Dose but received Vehicle instead)
Completed | 42 | 43 | 42
Not Completed | 1 | 1 | 0
Period: Safety Set (as Treated)
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle
Started | 42 (One subject was randomized to AXR-270 Low Dose but received Vehicle instead) | 43 (One subject withdrew consent and was withdrawn from the study prior to dosing with the assigned treatment because the subject was not able to comply with the visit schedule) | 43 (One subject was randomized to AXR-270 Low Dose but received Vehicle instead)
Completed | 41 | 42 | 43
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle | Total
Number analyzed (Participants) | 43 | 44 | 42 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.7) | 63.9 (17.4) | 64.3 (15.4) | 65.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 30 | 92
  Male | 9 | 16 | 12 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 38 | 37 | 115
  Black or African American | 2 | 2 | 3 | 7
  Asian | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 42 | 129
Total Meibomian Gland Dysfunction Score [Mean (Standard Deviation); unit: units on a scale] — The total MGD score is the sum of secretion of 5 central glands on the upper and lower eyelids. Each gland orifice was scored from 0-3. The total score range was from 0-15 per eyelid. The numbers reported are for the Study Eyelid of each subject (=eyelid with higher sum score of the Total MGD score and Vascularity of Eyelid Margin score at baseline). Lower scores indicate a better outcome.
  Scores: 0 = clear/slightly yellow; 1 = opaque/yellow, whitish, particulate; 2 = paste; 3 = none/occluded.
  units on a scale | 9.7 (1.6) | 9.5 (2.3) | 10.0 (2.3) | 9.7 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Incidence of treatment emergent ocular and systemic adverse events (TEAE)
Time Frame: 22 Days
Population: Safety Set
Measure: Number; unit: adverse events
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle
Number analyzed (Participants) | 42 | 43 | 43
adverse events
  Non-ocular TEAEs | 1 | 1 | 2
  Non-ocular Serious TEAEs | 0 | 0 | 0
  Ocular TEAEs | 0 | 0 | 4
  Ocular Serious TEAEs | 0 | 0 | 0

2. Secondary Outcome: Total Meibomian Gland Dysfunction Score
Description: Change from Baseline in total MGD score (Study Eyelid):
  The total MGD score is the sum of secretion of 5 central glands on the upper and lower eyelids. Each gland orifice was scored from 0-3. The total score range was from 0-15 per eyelid. The numbers reported are for the Study Eyelid of each subject (=eyelid with higher sum score of the Total MGD score and Vascularity of Eyelid Margin score at baseline). Greater negative scores indicate a better outcome.
  Scores: 0 = clear/slightly yellow; 1 = opaque/yellow, whitish, particulate; 2 = paste; 3 = none/occluded.
Time Frame: 22 Days
Population: Full Analysis Set (Intent-to-Treat)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle
Number analyzed (Participants) | 42 | 42 | 41
score on a scale | -0.9 (2.3) | -1.7 (2.1) | -2.1 (2.6)

ADVERSE EVENTS:
Time Frame: 22 days
Description: Treatment emergent ocular and non-ocular adverse events are based on the Safety Set
Arm/Group | AXR-270 Low Dose | AXR-270 High Dose | AXR-270 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 1/42 | 1/43 | 4/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXR-270 Low Dose (N=42) | AXR-270 High Dose (N=43) | AXR-270 Vehicle (N=43)
Covid (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
increased blood creatine phosphokinase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
mild urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
mild headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
mild eyelid pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
mild eyelid erythema, edema (Eye disorders) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement defined what qualifies as Confidential Information and restrictions on publication of study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT04469998/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04469998/SAP_001.pdf